CLINICAL TRIAL: NCT07113470
Title: Response to Combined Trigeminal and Occipital Nerve Stimulation for the Preventive Treatment in Chronic Cluster Headache: The RESPONSE-II Study
Brief Title: Response to Combined Trigeminal and Occipital Nerve Stimulation for the Preventive Treatment in Chronic Cluster Headache
Acronym: RESPONSE-II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salvia BioElectronics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SCI-04-CCH; NL-010395 (Other: CCMO)
Record Dates: First submitted 2025-07-29; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MySalvia Therapy (Experimental)
  Interventions: Device: The Salvia PRIMUS implantable neurostimulator System

INTERVENTIONS:
Device: The Salvia PRIMUS implantable neurostimulator System — The Salvia PRIMUS implantable neurostimulator System is designed to provide subcutaneous neurostimulation to the V1 branches of the Trigeminal nerves (supra-orbital and supra-trochlear nerves) and the branches of the Greater Occipital Nerves. It is intended to modulate headaches' neural networks by utilizing mild electrical pulses. There are 2 stimulation waveforms options: the Salvia burst waveform providing paresthesia-free stimulation and Tonic waveform, providing paresthesia-provoking stimulation. The PRIMUS System comprises a 25 cm (forehead) and a 17cm (back of the head) subcutaneous implant, a MySalvia device, a programmer, and surgical tooling.

SUMMARY:
This is a limited open-label study being performed at two centers in the Netherlands. All participants will receive the same treatment, and both the patients and doctors will know what that treatment is. The goal is to see how safe and effective the PRIMUS system is for preventing Chronic Cluster Headaches (CCH) in people who haven't responded well to the drug verapamil. The study will also look at the patients' experience using the system.

DETAILED DESCRIPTION:
During a Cluster Headache attack, the brain area called the hypothalamus may not do its usual job of blocking pain signals, which can make the pain worse. Stimulating the occipital nerves (at the back of the head) may help return brain activity in certain areas-like the hypothalamus, midbrain, and lower brainstem-back to normal. This could help reduce the brain's sensitivity to pain over time.

Stimulating another nerve group, called the V1 branch of the Trigeminal nerves (around the forehead and eye), can also help by interrupting pain signals and possibly stopping an attack or making it less severe and less frequent.

When both nerve areas-the Trigeminal and Occipital nerves-are stimulated together, it may have a stronger effect on reducing pain and how often headaches happen. Some early reports in a few patients have shown promising results with this combined treatment.

The PRIMUS system is a small device that can be implanted under the skin. It was designed to target both the Trigeminal and Occipital nerves at the same time, with a focus on treating severe head and face pain. It may offer relief for people with chronic cluster headaches who haven't been helped by medication.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent
2. 18 years of age or older
3. Documented Primary Chronic Cluster Headache, for at least 1 year as per ICHD-3 criteria

Exclusion Criteria:

1. Any other chronic primary or secondary headache disorder, unless they can clearly differentiate them from cluster headache attacks based on the quality and associated symptoms
2. Secondary Cluster Headache

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment | 12 weeks
  The primary safety assessment is the incidence of serious procedure and/or device-related adverse events in all subjects at the 12 week visit and at the end of the study. All adverse clinical events will be collected, coded and reported, throughout the duration of the study according to the definitions of ISO 14155:2020. Device and procedure-related adverse events will be distinguished from stimulation-related adverse events. All device deficiencies, as defined by ISO 14155:2020, will be documented and reported throughout the duration of the study.

IPD SHARING:
Plan to Share IPD: Undecided